CLINICAL TRIAL: NCT03831984
Title: Topical 0,09% Bromfenac for Intraoperative Miosis and Pain Reduction in Femtosecond Laser-assisted Cataract Surgery
Brief Title: Topical Bromfenac for Intraoperative Miosis and Pain Reduction
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Hospital de La Luz (Other)
Responsible Party: Principal Investigator, Maria Camila Aguilar Sierra, MD, Hospital de La Luz
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MAguilarSierra
Record Dates: First submitted 2019-02-04; First posted 2019-02-06 (Actual); Last update posted 2019-02-06 (Actual); Status verified 2019-02

CONDITIONS: Cataract
Keywords: Phacoemulsification; femtosecond laser; bromfenac; NSAID; pupil
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 0,09% Bromfenac (Active Comparator): Topical 0,09% Bromfenac twice daily 3 days before surgery
  Interventions: Drug: 0,09% Bromfenac
- 0,1% sodium hyaluronate (Placebo Comparator): Topical 0,1% sodium hyaluronate twice daily 3 days before surgery
  Interventions: Drug: 0,1% sodium hyaluronate

INTERVENTIONS:
Drug: 0,09% Bromfenac — topical 0,09% Bromfenac, one drop twice daily 3 days before surgery
  Other Names: Zebesten
  Arms: 0,09% Bromfenac
Drug: 0,1% sodium hyaluronate — topical 0,1% sodium hyaluronate, one drop twice daily 3 days before surgery
  Other Names: Hyabak
  Arms: 0,1% sodium hyaluronate

SUMMARY:
To evaluate the effect of bromfenac ophthalmic solution 0.09% for reduction of intraoperative miosis and pain in patient who have undergone femtosecond laser-assisted cataract surgery.

DETAILED DESCRIPTION:
This prospective cross-sectional randomized clinical study included 60 patients with senile cataract in the absence of significant ocular comorbidity. The patients received 0.09% bromfenac ophthalmic solution or control placebo twice a day for 3 days before surgery. Pupil diameter was measured at the initiation and finalization of femtosecond laser-assisted cataract surgery and pain quantification was assessed by analogous pain scale at one day follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Male and female
* Subjects 18 years or older
* Patients scheduled for unilateral femtosecond laser-assisted cataract surgery cataract surgery with posterior chamber (PC) IOL implantation.

Exclusion Criteria:

* Presence of corneal abnormalities
* History of intraocular surgery
* History of ocular or systematic diseases (glaucoma, diabetes, uveitis
* Regular, systemic use of steroid or NSAIDs during the previous 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2018-11-30 (Actual); Study Completion 2019-03-30 (Estimated)

PRIMARY OUTCOMES:
intraoperative miosis | 2 days
  Evaluation of reduction of intraoperative miosis before and after femtosecond laser assisted cataract surgery

SECONDARY OUTCOMES:
postoperative pain | 1 day
  Evaluation of reduction of postoperative pain using a visual analogue scale

CONTACTS AND LOCATIONS:
Overall Officials: MARIA AGUILAR SIERRA, MD, Principal Investigator — FELLOWSHIP
Locations (1):
- Maria Camila Aguilar Sierra, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No